CLINICAL TRIAL: NCT06122415
Title: The Swedish BioFINDER - Memory Clinic Study
Acronym: Validate
Status: Recruiting | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Erik Stomrud, M.D., PhD, Skane University Hospital
Other Study IDs: Validate
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Mild Dementia; Mild Cognitive Impairment; SCD; Alzheimer Disease; Lewy Body Disease; Frontotemporal Degeneration; Vascular Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients in secondary care with cognitive symptoms
  Interventions: Diagnostic Test: Plasma Amyloid Probability Score 2 (APS 2) score; Diagnostic Test: Plasma ptau217/nptau217; Diagnostic Test: Plasma ptau217; Diagnostic Test: Plasma neurofilament light (NfL); Diagnostic Test: Plasma Ab42/Ab40

INTERVENTIONS:
Diagnostic Test: Plasma Amyloid Probability Score 2 (APS 2) score — APS 2 score (combination of ptau217/nptau217 and Ab42/Ab40). The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma ptau217/nptau217 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma ptau217 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma neurofilament light (NfL) — The cut off will be predefined. The samples will be analysed prospectively every two weeks.
Diagnostic Test: Plasma Ab42/Ab40 — The cut off will be predefined. The samples will be analysed prospectively every two weeks.

SUMMARY:
The diagnosis of diseases causing memory difficulties or dementia is often challenging. Without the use of advanced methods such as cerebrospinal fluid tests, approximately 25-30% do not receive a correct diagnosis today. However, the investigators have recently developed new blood biomarkers with high diagnostic accuracy, and the investigators now want to investigate whether they can eventually replace cerebrospinal fluid tests. This is because blood tests are much more cost-effective and significantly easier for patients compared to cerebrospinal fluid tests.

In this study, 1200 patients undergoing clinical evaluations at the Memory Clinic, Skåne University Hospital in Malmö, are included for blood and cerebrospinal fluid sample collection. The blood samples are sent for analysis using the new blood biomarkers. Subsequently, the results are compared with those from the clinical analysis of cerebrospinal fluid to determine how well they perform in routine clinical practice as an alternative to cerebrospinal fluid tests and whether the blood test improves patient care. This comparison is carried out by the attending physician in three steps:

1. Assessment without access to the results of either the blood test or cerebrospinal fluid test.
2. Assessment with access to only the results of the blood test.
3. Assessment with access to the results of both the blood test and cerebrospinal fluid test.

Aim 1) To prospectively validate plasma Alzheimer's disease (AD) biomarkers for diagnosis of patients with cognitive symptoms who are evaluated in a specialist memory clinic.

Aim 2) Determine whether blood AD biomarkers improve patient management in specialist memory clinic settings.

DETAILED DESCRIPTION:
The diagnosis of diseases causing memory difficulties or dementia is often challenging. Without the use of advanced methods such as cerebrospinal fluid tests, approximately 25-30% do not receive a correct diagnosis today. However, the investigators have recently developed new blood biomarkers with high diagnostic accuracy, and the investigators now want to investigate whether they can eventually replace cerebrospinal fluid tests. This is because blood tests are much more cost-effective and significantly easier for patients compared to cerebrospinal fluid tests.

In this study, 1200 patients undergoing clinical evaluations at the Memory Clinic, Skåne University Hospital in Malmö, are included for blood and cerebrospinal fluid sample collection. The blood samples are sent for analysis using the new blood biomarkers. Subsequently, the results are compared with those from the clinical analysis of cerebrospinal fluid to determine how well they perform in routine clinical practice as an alternative to cerebrospinal fluid tests and whether the blood test improves patient care. This comparison is carried out by the attending physician in three steps:

1. Assessment without access to the results of either the blood test or cerebrospinal fluid test.
2. Assessment with access to only the results of the blood test.
3. Assessment with access to the results of both the blood test and cerebrospinal fluid test.

Aim 1) To prospectively validate plasma AD biomarkers for diagnosis of patients with cognitive symptoms who are evaluated in a specialist memory clinic. The investigators here intend to study the clinical robustness and accuracy of plasma AD biomarkers in real-world settings by using high-performing plasma assays over 2-3 years, focusing on a specialist memory clinic population (n=1200). In this study plasma samples are collected as part of clinical praxis and analyzed on a bi-weekly basis throughout the study period (and not in single batches/at study closure). The investigators will (1) use pre-defined cut offs for each biomarker (similar to real world clinical practice), and (2) use an accurate reference standard (i.e., presence of AD brain pathology as determined with cerebrospinal fluid (CSF) Aβ42/Aβ40 [Lumipulse; Fujirebio] and CSF P-tau217 [Eli Lilly]). The investigators will strive to recruit diverse and representative populations of patients with subjective cognitive decline (SCD), mild cognitive impairment (MCI) and mild dementia. The effects of potential confounders (such as kidney function) on diagnostic accuracy will also be studied. The investigators will only use really top-performing plasma assays for each biomarker, including p-tau217 and Ab42/Ab40.

Expected outcomes: The investigators will 1) determine the diagnostic accuracy of different plasma AD biomarkers, 2) establish an optimal combination of plasma biomarkers for detection of AD brain pathology and 3) identify the effects of different potential confounding factors (e.g., kidney function) on the performance of different plasma biomarkers, when used prospectively in both real-world specialist and primary care populations.

Aim 2) Determine whether blood AD biomarkers improve patient management in specialist memory clinic settings. As often noted by regulatory authorities, it is important to know if novel diagnostic methods improve the actual management of patients in real world settings. Consequently, the investigators study whether the most promising plasma biomarkers for symptomatic AD (including plasma p-tau217) will improve AD diagnosis beyond what is currently done as part of clinical practice. The dementia experts will document the most likely diagnosis (and the certainty of the diagnosis) after having performed an interview with the patient and informant, as well as evaluated the patient's cognitive test results, routine blood tests and structural brain imaging. The physician will then re-evaluate the diagnosis (and certainty of diagnosis) after having obtained the plasma p-tau217 results, and the pre- and posttest diagnosis will be compared to the reference standard (i.e., presence of AD brain pathology as determined with CSF Aβ42/Aβ40 [Lumipulse; Fujirebio] and CSF P-tau217 [Eli Lilly]). Change in treatment and care of the patient after evaluating the p-tau217 results will also be recorded similar to how amyloid-positron emission tomography (PET) was evaluated in the IDEAS study.

Expected outcomes: The investigators will determine whether the addition of plasma AD biomarkers to current clinical practice in memory clinics and/or primary care improves diagnosis and management of patients with SCD, MCI or mild dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Under investigation for cognitive symptoms at the Memory clinic.
2. Cerebrospinal fluid and blood sampling is planned to be done as part of clinical practice even if the patient is not taking part of this study.

Exclusion Criteria:

1. Not undergoing CSF or blood sampling as part of clinical practice.
2. Not undergoing cognitive testing as part of clinical practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cognitive symptoms (SCD, MCI or dementia) at a secondary memory clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain AD pathology as determined by CSF AD biomarkers | At baseline (cross-sectional)
  CSF Ab42/Ab40 and p-tau217

SECONDARY OUTCOMES:
Clinical diagnosis supported by CSF biomarkers | At baseline (cross-sectional)
  Clinical diagnosis based on The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) but supported by CSF biomarkers
Brain AD pathology as determined by amyloid amyloid PET imaging | At baseline (cross-sectional)
  Amyloid PET imaging
Brain AD pathology as determined by tau PET imaging | At baseline (cross-sectional)
  Tau PET imaging
Progression to AD dementia in patients with SCD or MCI at baseline | At baseline (cross-sectional)
  Development of AD dementia during follow-up diagnosed using DSM-5 and supported by CSF biomarkers
Change in patient management | At baseline (cross-sectional)
  Change in suggested diagnosis, treatment, referral or ordered diagnostic tests
Change in diagnostic confidence | At baseline (cross-sectional)
  Change in diagnostic confidence of the treating physician

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year after study completion